CLINICAL TRIAL: NCT00464620
Title: A Phase II Trial of Dasatinib in Advanced Sarcomas
Brief Title: Trial of Dasatinib in Advanced Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC009
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-10

CONDITIONS: Rhabdomyosarcoma; Malignant Peripheral Nerve Sheath Tumors; Chondrosarcoma; Sarcoma, Ewing's; Sarcoma, Alveolar Soft Part; Chordoma; Epithelioid Sarcoma; Giant Cell Tumor of Bone; Hemangiopericytoma; Gastrointestinal Stromal Tumor (GIST)
Keywords: Dasatinib; Rhabdomyosarcoma; Malignant peripheral nerve sheath tumor; Chondrosarcoma; Ewing's; Alveolar soft part sarcoma (ASPS); Chordoma; Epithelioid sarcoma; Giant cell tumor of bone; Hemangiopericytoma/solitary fibrous tumor; Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Rhabdomyosarcoma; Neurofibrosarcoma; Chondrosarcoma; Sarcoma, Ewing; Sarcoma, Alveolar Soft Part; Chordoma; Sarcoma; Giant Cell Tumor of Bone; Hemangiopericytoma; Gastrointestinal Stromal Tumors; Solitary Fibrous Tumors | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib, 70 mg, twice daily (Experimental): Patients take 70 mg of Dasatinib, twice daily, for 28 day cycles
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — oral agent, continuous dosing, Cycles = 28 days

SUMMARY:
This study will examine the response rate and the 6-month progression-free survival rates of subjects with advanced sarcoma treated with dasatinib.

DETAILED DESCRIPTION:
Further details provided by SARC (Sarcoma Alliance for Research through Collaboration):

Treatment: Subjects take Dasatinib twice daily by mouth for 28 days per 28 day cycle.

Subjects will be seen for interim medical history, physical exam and laboratory studies prior to each cycle. Subjects will undergo tumor imaging every 2 months (8 weeks) for the first 6 months and approximately every 3 months thereafter while on treatment.

A blood sample for collection of specimens with which to later study serum level of Dasatinib and effects on biomarkers of drug activity will be obtained approximately 2 to 4 weeks after the start of treatment.

Central collection of archival tumor with which to later study the frequency of expression and/or mutation of kinases inhibited by dasatinib will occur.

Subjects will be followed for approximately every 3 months until 2 years from registration and then approximately yearly until 5 years from registration.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable, recurrent, or metastatic histologically-confirmed soft tissue or bone sarcoma of one of the following subtypes:

   * Leiomyosarcoma --* NO LONGER ELIGIBLE*
   * Liposarcoma--* NO LONGER ELIGIBLE*
   * Malignant fibrous histiocytoma (MFH)/pleomorphic undifferentiated sarcoma--* NO LONGER ELIGIBLE*
   * Rhabdomyosarcoma --* NO LONGER ELIGIBLE*
   * Malignant peripheral nerve sheath tumor (MPNST) --* NO LONGER ELIGIBLE*
   * Osteosarcoma (skeletal or extraosseous)--* NO LONGER ELIGIBLE*
   * Ewing's --* NO LONGER ELIGIBLE*
   * Chondrosarcoma
   * Alveolar soft part sarcoma
   * Chordoma
   * Epithelioid sarcoma
   * Giant cell tumor of bone
   * Hemangiopericytoma/solitary fibrous tumor
   * Gastrointestinal Stromal Tumor (GIST) --* NO LONGER ELIGIBLE*
2. Documentation that subjects with leiomyosarcoma, liposarcoma, osteosarcoma, Ewing's, MPNST, rhabdomyosarcoma or MFH have received, not been eligible for or refused at least one prior chemotherapy regimen before participation in the dasatinib study. Subjects with GIST must have received or been intolerant to imatinib; prior treatment with other agents including sunitinib is not required.Neoadjuvant/adjuvant chemotherapy qualifies as prior therapy.
3. Subjects must have unidimensionally measurable lesion(s) either by x-ray, computed tomography (CT), magnetic resonance imaging (MRI) or physical examination documented within 30 days prior to registration.
4. Prior radiation will be allowed. More than two weeks should have elapsed since the administration of the last fraction of radiation therapy, and subjects must have recovered from grade 2 or higher associated toxicities. Measurable lesions, which are selected as target lesions, must be outside previously radiated fields or have documented progression no sooner than 6 weeks after completion of radiation.
5. More than 2 weeks must have elapsed since the subject has received any prior systemic chemotherapy (6 weeks for mitomycin C), and the patient should have recovered from toxicities to the baseline prior to the last course of chemotherapy.
6. Adequate hematologic function within 14 days prior to registration.
7. Prothrombin Time (PT) (or INR) and Partial Thromboplastin Time (PTT) ≤ 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to registration.
8. Serum creatinine ≤ 2.0 times the institutional ULN within 14 days prior to registration.
9. Serum magnesium, potassium and adjusted (or ionized) calcium ≥ the institutional lower limit of normal (LLN). (Supplementation of electrolytes prior to screening is allowed).
10. Left ventricular ejection fraction ≥ 45% measured by echocardiogram or multiple gated acquisition (MUGA) within 30 days prior to registration (but must be performed after the last dose of an anthracycline) for subjects who have received an anthracycline (e.g. doxorubicin, epirubicin) or have a medical history of cardiac disease. The measurement of left ventricular ejection fraction is not required of subjects whom have not received cardiotoxic chemotherapy (e.g. anthracycline) and do not have a medical history of cardiac disease.
11. Sexually active women and men of childbearing potential must agree to use an effective method of birth control during the course of the study and for up to 3 months following the last dose of the study drug, in a manner such that risk of pregnancy is minimized. Surgical sterilization, intrauterine device or barrier method (e.g. condom and/or diaphragm with spermicidal agents) are acceptable forms of birth control.
12. Women of childbearing potential must have a negative pregnancy test (urine or serum) within 7 days prior to treatment. A pregnancy test is not required for registration. Women who have not menstruated for more than 2 years will be considered postmenopausal, thus not of childbearing potential.
13. Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2.
14. Weight ≥ 50 kg because there is limited experience with dasatinib in subjects weighing less than 50 kg.
15. ≥13 years of age Minors will be required to sign an assent document prior to treatment.
16. Subjects must be able to swallow whole tablets.
17. Subjects must be informed of the investigational nature of the study and provide written, informed consent and authorization to release protected health information using a document(s) approved by the investigator's institution.
18. A paraffin block, either from a previous surgery or recent biopsy, should be available for correlative studies. If a block of tumor is not available, at least 8 unstained slides of tumor sample, 1 H&E and three (3) 15 micron-thick sections in an eppendorf tube for DNA extraction from a representative portion of the sarcoma may be substituted after discussion with and approval from the study Principal Investigator.

Exclusion Criteria:

1. Subjects who are curable by conventional multidisciplinary management.
2. Subjects with symptomatic central nervous system metastasis.
3. Women who are pregnant or nursing/breastfeeding.
4. History of significant bleeding disorder unrelated to cancer, including:

   * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
   * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
5. Subjects currently taking medications that inhibit platelet function (i.e., aspirin, dipyridamole, epoprostenol, eptifibatide, clopidogrel, cilostazol, abciximab, ticlopidine, and any non-steroidal anti-inflammatory drug) because of a potential increased risk of bleeding from dasatinib.
6. Subjects currently taking anticoagulants (warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, enoxaparin]) because of a potential increased risk of bleeding from dasatinib.
7. Diagnosis of unstable angina or myocardial infarction within 6 months of study entry.
8. Subjects currently taking one or more of the following drugs that are generally accepted to have a risk of causing Torsades de Pointes:

   * Quinidine, procainamide, disopyramide
   * Amiodarone, sotalol, ibutilide, dofetilide
   * Erythromycins, clarithromycin
   * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
   * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.
9. Diagnosed or suspected congenital long QT syndrome.
10. Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec) within 30 days prior to study registration.
11. Subjects unable or unwilling to suspend treatment with bisphosphonates for at least the first 8 weeks of treatment with study drug because of the risk of hypocalcemia caused by dasatinib.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2007-05; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, MD, PhD, Principal Investigator — University of Michigan
Locations (20):
- United States (20):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Kootenai Cancer Center, Coeur d'Alene, Idaho
  - Oncology Specialists, Park Ridge, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson, Houston, Texas

REFERENCES:
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients with GIST were enrolled between June 2008 and December 2009 and 48 were evaluable for response. Between May 2007 and May 2009, 200 patients with advanced, high-grade sarcoma were enrolled into the aggressive subtype for this study. 116 patients were registered beginning in July 2007 to the indolent subtype for this study.
Groups:
- GIST: Dasatinib, 70 mg, Twice Daily; Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily; Indolent Subtype: Dasatinib, 70 mg, Twice Daily: Patients take 70 mg of Dasatinib, twice daily, for 28 day cycles
  Dasatinib: oral agent, continuous dosing, Cycles = 28 days
Period: Overall Study
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Started | 50 | 200 | 116
Completed | 48 (48 patients were evaluable.) | 198 | 109
Not Completed | 2 | 2 | 7
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Ineligible sarcoma subtype | 0 | 2 | 2
Not completed — Use of prohibited concomitant medication | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: 116 subjects enrolled in the Indolent subtype, however 109 subjects began treatment. Baseline characteristics for the Indolent subtype were based off of 109 subjects on treatment. This explains the discrepancy between the Participant Flow and the Overall Number of Baseline Participants.
Arm/Group | Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 359
Age, Continuous [Median (Full Range); unit: years] — Population: The baseline measurements are categorized by the three different subtypes from the protocol (aggressive, indolent and GIST).
  years
    Aggressive subtype: number analyzed (Participants) | 200
    Aggressive subtype | 52 [14.8 to 87.3]
    GIST: number analyzed (Participants) | 50
    GIST | 60 [19 to 78]
    Indolent: number analyzed (Participants) | 109
    Indolent | 54 [22 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The baseline measurements are categorized by the three different subtypes from the protocol (aggressive, indolent and GIST).
  Participants
    Aggressive subtype: number analyzed (Participants) | 200
    Aggressive subtype: Female | 96
    Aggressive subtype: Male | 104
    GIST: number analyzed (Participants) | 50
    GIST: Female | 19
    GIST: Male | 31
    Indolent: number analyzed (Participants) | 109
    Indolent: Female | 33
    Indolent: Male | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The baseline measurements are categorized by the three different subtypes from the protocol (aggressive, indolent and GIST).
  Participants
    Aggressive subtype: number analyzed (Participants) | 200
    Aggressive subtype: White | 171
    Aggressive subtype: Black | 15
    Aggressive subtype: Asian | 6
    Aggressive subtype: Other | 6
    Aggressive subtype: Unknown | 2
    Aggressive subtype: Native American | 0
    GIST: number analyzed (Participants) | 50
    GIST: White | 41
    GIST: Black | 3
    GIST: Asian | 3
    GIST: Other | 1
    GIST: Unknown | 1
    GIST: Native American | 1
    Indolent: number analyzed (Participants) | 109
    Indolent: White | 94
    Indolent: Black | 8
    Indolent: Asian | 3
    Indolent: Other | 4
    Indolent: Unknown | 0
    Indolent: Native American | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate: Number of Participants With Objective Tumor Response
Description: Assessment of objective tumor response for response rate with MRI or CT using Choi criteria: Complete Remission (CR) Complete disappearance of all measurable and evaluable disease for at least 4 weeks; Partial Remission (PR) A 10% or greater decrease from the baseline in the sum of the largest diameters of all measurable target lesions.
Time Frame: Up to 24 months
Population: 116 subjects enrolled in the Indolent subtype, however 109 subjects began treatment. 50 patients enrolled in the GIST subtype, however 48 patients were evaluable. This explains the discrepancy between Overall Number of Participants Analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 48 | 198 | 109
Participants | 12 | 14 | 20

2. Primary Outcome: 6 Month Progression-free Survival Rate of "Indolent" Sarcomas Treated With Dasatinib
Description: Estimate the 6 month progression-free survival rate of "indolent" sarcomas treated with dasatinib. Progression is defined using Choi criteria, as a 10% or greater increase in the sum of all measurable target lesions over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or unequivocal reappearance of any lesion which had disappeared, or appearance of any new lesions of greater than double slice thickness in size, or any new or enlarging solid nodule in a previously hypodense treated mass.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Indolent Subtypes: Dasatinib, 70 mg, Twice Daily: Patients take 70 mg of Dasatinib, twice daily, for 28 day cycles
  Dasatinib: oral agent, continuous dosing, Cycles = 28 days
Arm/Group | Indolent Subtypes: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 109
Participants | 52

3. Primary Outcome: 6 Month Progression-free Survival Rate of Gastrointestinal Stromal Tumors (GIST)
Description: To estimate the 6 month progression-free survival rate of gastrointestinal stromal tumors (GIST). Progression is defined using Choi criteria, as a 10% or greater increase in the sum of all measurable target lesions over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, or clear worsening of any evaluable disease, or unequivocal reappearance of any lesion which had disappeared, or appearance of any new lesions of greater than double slice thickness in size, or any new or enlarging solid nodule in a previously hypodense treated mass.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 48
Participants | 14

4. Secondary Outcome: Median Time-to-progression of Subjects With GIST Treated With Dasatinib.
Description: To estimate the median time-to-progression of subjects with GIST treated with dasatinib.
Time Frame: Up to 30 months
Measure: Median (Full Range); unit: months
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 48
months | 2.9 [2 to 5.5]

5. Secondary Outcome: Overall Survival Rates at 2 and 5 Years From Registration of Subjects Treated With Dasatinib.
Description: To estimate the overall survival rates at 2 and 5 years from registration of subjects treated with dasatinib.
Time Frame: At 2 and 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 48 | 109
Participants
  2 years overall survival | 21 | 48
  5 years overall survival | 8 | 14

6. Secondary Outcome: Median Time-to-progression of Subjects With "Indolent" Sarcomas Treated With Dasatinib.
Description: To estimate the median time-to-progression of subjects with "indolent" sarcomas treated with dasatinib.
Time Frame: Up to 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 109
months | 5.8 [3.7 to 7.4]

7. Secondary Outcome: 6 Month Progression-free Survival Rate of Subjects Enrolled in the Aggressive Subtype.
Description: To estimate the 6 month progression-free survival rate of subjects with leiomyosarcoma, liposarcoma, osteosarcoma including high-grade chondrosarcomas, Ewing's sarcoma, Malignant fibrous histiocytoma (MFH), rhabdomyosarcoma and MPNST treated with dasatinib.
Time Frame: At 6 months
Population: The numbers analyzed in one or more rows are different because they are broken up by cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 198
Participants
  UPS: number analyzed (Participants) | 48
  UPS | 6
  Leiomyosarcoma: number analyzed (Participants) | 49
  Leiomyosarcoma | 5
  Osteosarcoma: number analyzed (Participants) | 46
  Osteosarcoma | 5
  Rhabdomyosarcoma: number analyzed (Participants) | 13
  Rhabdomyosarcoma | 0
  Ewing's Sarcoma: number analyzed (Participants) | 17
  Ewing's Sarcoma | 1
  Liposarcoma: number analyzed (Participants) | 11
  Liposarcoma | 0
  MPNST: number analyzed (Participants) | 14
  MPNST | 0

8. Secondary Outcome: Median Time-to-progression of Subjects Enrolled in the Aggressive Subtype.
Description: To estimate the median time-to-progression of subjects with leiomyosarcoma, liposarcoma, osteosarcoma including high-grade chondrosarcomas, Ewing's sarcoma, MFH, rhabdomyosarcoma and MPNST treated with dasatinib.
Time Frame: Up to 37 weeks
Measure: Median (Full Range); unit: months
Arm/Group | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 198
months | 1.9 [0.9 to 2.2]

9. Secondary Outcome: Overall Survival Rates at 2 and 5 Years From Registration of Subjects Enrolled in the Aggressive Subtype Treated With Dasatinib.
Description: To estimate the overall survival rates at 2 and 5 years from registration of subjects enrolled in the aggressive subtype treated with dasatinib.
Time Frame: At 2 and 5 years
Population: The number analyzed in one or more rows differs from overall number because the rows are broken down into cohorts. The counts in the categories will not add up to the number analyzed, because those numbers represent number of participants that have reached overall survival at 2 and 5 years.
Measure: Number; unit: participants
Arm/Group | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 198
participants
  Ewing's Sarcoma : 2 year overall survival rate: number analyzed (Participants) | 17
  Ewing's Sarcoma : 2 year overall survival rate | 7
  Ewing's Sarcoma : 5 year overall survival rate: number analyzed (Participants) | 7
  Ewing's Sarcoma : 5 year overall survival rate | 0
  Leiomyosarcoma : 2 year overall survival rate: number analyzed (Participants) | 49
  Leiomyosarcoma : 2 year overall survival rate | 21
  Leiomyosarcoma : 5 year overall survival rate: number analyzed (Participants) | 21
  Leiomyosarcoma : 5 year overall survival rate | 2
  Liposarcoma : 2 year overall survival rate: number analyzed (Participants) | 11
  Liposarcoma : 2 year overall survival rate | 0
  Liposarcoma : 5 year overall survival rate: number analyzed (Participants) | 11
  Liposarcoma : 5 year overall survival rate | 0
  MPNST : 2 year overall survival rate: number analyzed (Participants) | 14
  MPNST : 2 year overall survival rate | 0
  MPNST : 5 year overall survival rate: number analyzed (Participants) | 14
  MPNST : 5 year overall survival rate | 0
  Osteosarcoma : 2 year overall survival rate: number analyzed (Participants) | 46
  Osteosarcoma : 2 year overall survival rate | 15
  Osteosarcoma : 5 year overall survival rate: number analyzed (Participants) | 15
  Osteosarcoma : 5 year overall survival rate | 0
  Rhabdomyosarcoma : 2 year overall survival rate: number analyzed (Participants) | 13
  Rhabdomyosarcoma : 2 year overall survival rate | 8
  Rhabdomyosarcoma : 5 year overall survival rate: number analyzed (Participants) | 8
  Rhabdomyosarcoma : 5 year overall survival rate | 7
  UPS : 2 year overall survival rate: number analyzed (Participants) | 48
  UPS : 2 year overall survival rate | 26
  UPS : 5 year overall survival rate: number analyzed (Participants) | 26
  UPS : 5 year overall survival rate | 6

10. Secondary Outcome: Uni-dimensional and Bi-dimensional Tumor Size, Tumor Volumes and Tumor Average Density Determined by Computer-aided Automated Detection in a Subset of Subjects With Tumor Predominately Involving the Lung
Description: To prospectively collect uni-dimensional and bi-dimensional tumor size, tumor volumes and tumor average density determined by computer-aided automated detection in a subset of subjects with tumor predominately involving the lung
Time Frame: Up to 37 weeks
Population: This data was not collected because the imaging software and work station was not obtained.
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Plasma Level of Dasatinib and Inhibition of SRC and/or Focal Adhesion Kinase (FAK) in Peripheral Blood Mononuclear Cells
Description: Obtain blood samples to characterize plasma level of dasatinib and inhibition of SRC and/or FAK in peripheral blood mononuclear cells 2 hours after ingestion of drug at 2-4 weeks from the start of treatment if activity of the drug in a sarcoma subtype warrants further study.
Time Frame: 2-4 weeks from start of treatment
Population: Evaluation of blood levels of drug was not performed because there was insufficient activity and the level of activity did not warrant further study.
Arm/Group | GIST: Dasatinib, 70 mg, Twice Daily | Aggressive Subtypes: Dasatinib, 70 mg, Twice Daily | Indolent Subtype: Dasatinib, 70 mg, Twice Daily
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Tumors With Kinase Expression
Description: Obtain tumor tissue for creation of tissue microarrays to examine the frequency of kinase expression such as SRC and/or FAK in leiomyosarcoma, liposarcoma, osteosarcoma, MFH, rhabdomyosarcoma, MPNST, chondrosarcoma, Ewing's, Alveolar soft part sarcoma (ASPS), chordoma, epithelioid sarcoma, giant cell tumor of bone, hemangiopericytoma, and GIST if activity of the drug in a subtype warrants further study. The outcome measure demonstrates the number of participants who had tissue that was able to generate tissue microarray for kinase expression.
Time Frame: Up to 37 weeks
Population: The overall number of participants analyzed demonstrates the number of participants whose tumor samples received. The results illustrate the tissue that was able to generate tissue microarray for SRC and FAK analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Osteosarcoma; Leiomyosarcoma; MFH/Undifferentiated Pleomorphic Sarcoma: Patients take 70 mg of Dasatinib, twice daily, for 28 day cycles
  Dasatinib: oral agent, continuous dosing, Cycles = 28 days
Arm/Group | Osteosarcoma | Leiomyosarcoma | MFH/Undifferentiated Pleomorphic Sarcoma
Number analyzed (Participants) | 32 | 44 | 37
Participants | 11 | 24 | 16

13. Secondary Outcome: Number of Participants With Tumors With Mutations in Kinases
Description: Obtain tumor tissue to examine the frequency of mutations in kinases such as PDGFR in leiomyosarcoma, liposarcoma, osteosarcoma, MFH, rhabdomyosarcoma, MPNST, chondrosarcoma, Ewing's, ASPS, chordoma, epithelioid sarcoma, giant cell tumor of bone, hemangiopericytoma and GIST if activity of the drug in a subtype warrants further study. The outcome measure demonstrates the tissue that was able to generate tissue microarray for PDGFR analysis.
Time Frame: Up to 37 weeks
Population: The overall number of participants analyzed demonstrates the number of participants whose tumor samples were received. The results illustrate the tissue that was able to generate tissue microarray for PDGFR analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Osteosarcoma | Leiomyosarcoma | MFH/Undifferentiated Pleomorphic Sarcoma
Number analyzed (Participants) | 32 | 44 | 37
Participants | 11 | 24 | 16

ADVERSE EVENTS:
Groups:
- GIST, Aggressive, Indolent Subtypes: Patients take 70 mg of Dasatinib, twice daily, for 28 day cycles
  Dasatinib: oral agent, continuous dosing, Cycles = 28 days
Arm/Group | GIST, Aggressive, Indolent Subtypes
Serious Adverse Events (participants affected / at risk) | 158/355
Other Adverse Events (participants affected / at risk) | 314/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIST, Aggressive, Indolent Subtypes (N=355)
Allergic reaction (Immune system disorders) | 1 (1)
ALT (Investigations) | 2 (4)
Amylase (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AST (Investigations) | 2 (2)
Bilirubin (Investigations) | 1 (1)
Blood-other (Blood and lymphatic system disorders) | 1 (1)
CNS hemorrhage (Nervous system disorders) | 4 (4)
Coagulation-other (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4)
Confusion (Psychiatric disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4)
Constitutional symptoms-other (General disorders) | 1 (1)
Creatinine (Investigations) | 5 (5)
Death, NOS (General disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 11 (11)
Dermatology- other (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (11)
Disease progression, NOS (General disorders) | 7 (7)
Distention (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 34 (37)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 15 (16)
Flu-like syndrome (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
GI Hemorrhage: lower GI (Gastrointestinal disorders) | 2 (2)
GI Hemorrhage: upper GI (Gastrointestinal disorders) | 2 (2)
GI Obstruction: small bowel (Gastrointestinal disorders) | 6 (6)
GI Obstruction: stomach (Gastrointestinal disorders) | 1 (1)
GI Pain: abdomen (Gastrointestinal disorders) | 12 (12)
GI Ulcer: colon (Gastrointestinal disorders) | 1 (1)
GI- other (Gastrointestinal disorders) | 1 (1)
GU Hemorrhage: urinary (Renal and urinary disorders) | 2 (2)
GU Hemorrhage: vagina (Renal and urinary disorders) | 1 (1)
GU Infection, 0-2 ANC: urinary tract (Renal and urinary disorders) | 1 (1)
GU Infection, Unk ANC: ureter (Renal and urinary disorders) | 1 (1)
GU Pain: kidney (Renal and urinary disorders) | 1 (1)
Hemoglobin (Investigations) | 14 (15)
Hemorrhage-other (General disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Infection, Unk ANC: blood (Infections and infestations) | 2 (2)
Infection-other (Infections and infestations) | 5 (6)
Leukocytes (Investigations) | 1 (1)
Lung infection, 0-2 ANC: bronchus (Infections and infestations) | 1 (1)
Lung Infection, 3-4 ANC: bronchus (Infections and infestations) | 1 (1)
Lung Infection, Unk ANC: lung (Infections and infestations) | 1 (1)
Lung Pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Anxiety (Psychiatric disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Musculo. Pain (Musculoskeletal and connective tissue disorders) | 17 (17)
Nausea (Gastrointestinal disorders) | 18 (20)
Neuropathy- sensory (Nervous system disorders) | 1 (1)
Neutrophils (Investigations) | 2 (2)
Pain (General disorders) | 5 (5)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelets (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 30 (34)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary-other (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 5 (5)
Seizure (Nervous system disorders) | 1 (1)
Reproductive pain: pelvis (Reproductive system and breast disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 6 (6)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (19)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Sweating (Vascular disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (7)
Lymphopenia (Investigations) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
GI Hemorrhage- abdomen (Gastrointestinal disorders) | 1 (1)
GI Hemorrhage- esophagus (Gastrointestinal disorders) | 1 (1)
GI Hemorrhage- rectum (Gastrointestinal disorders) | 2 (2)
GI Hemorrhage- stomach (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema- limb (General disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Gait/walking (General disorders) | 1 (1)
Myelitis (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Pelvis pain (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GIST, Aggressive, Indolent Subtypes (N=355)
Anorexia (Metabolism and nutrition disorders) | 45 (49)
Constipation (Gastrointestinal disorders) | 27 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 45 (55)
Diarrhea (Gastrointestinal disorders) | 73 (99)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 56 (78)
Edema (General disorders) | 34 (50)
Fatigue (General disorders) | 113 (144)
Fever (General disorders) | 27 (29)
Hyperglycemia (Metabolism and nutrition disorders) | 25 (41)
Nausea (Gastrointestinal disorders) | 81 (93)
Pain- Other (General disorders) | 17 (17)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 43 (60)
Rash (Skin and subcutaneous tissue disorders) | 52 (64)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (31)
Vomiting (Gastrointestinal disorders) | 36 (38)
GI Pain: abdomen (Gastrointestinal disorders) | 15 (22)
Anemia (Blood and lymphatic system disorders) | 70 (103)
Hyponatremia (Metabolism and nutrition disorders) | 14 (18)
Headache (Nervous system disorders) | 52 (68)
Rigors/chills (General disorders) | 16 (18)
Weight loss (Investigations) | 17 (17)
Palpaitations (Cardiac disorders) | 2 (2)
Prolonged QTc (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 4 (4)
Hypertension (Vascular disorders) | 5 (6)
Cardiac- Other (Cardiac disorders) | 4 (5)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Elevated PTT (Investigations) | 3 (4)
Auditory/Ear- Other (Ear and labyrinth disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (4)
Dry eye (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Ocular- Other (Eye disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 8 (8)
Sweating (Vascular disorders) | 8 (9)
Heartburn (Gastrointestinal disorders) | 9 (10)
Distention (Gastrointestinal disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Taste alteration (Gastrointestinal disorders) | 8 (8)
Gastritis (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (6)
Hemorrhoids (Gastrointestinal disorders) | 6 (9)
Gastrointestinal- Other (Gastrointestinal disorders) | 7 (7)
Mucositis (Gastrointestinal disorders) | 4 (4)
Fistula (Gastrointestinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urine color change (Renal and urinary disorders) | 1 (1)
Bladder spasms (Renal and urinary disorders) | 2 (2)
Renal - Other (Renal and urinary disorders) | 5 (5)
Ureter obstruction (Renal and urinary disorders) | 1 (1)
Leukopenia (Investigations) | 13 (19)
Neutropenia (Investigations) | 15 (28)
Lymphopenia (Investigations) | 11 (12)
CNS Hemorrhage (Nervous system disorders) | 2 (2)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
GI Hemorrhage (Gastrointestinal disorders) | 9 (10)
GU Hemorrhage (Renal and urinary disorders) | 3 (5)
Lung Infection (Infections and infestations) | 14 (16)
GU Infection (Infections and infestations) | 4 (4)
Allergic reaction (Immune system disorders) | 1 (1)
GI Infection (Infections and infestations) | 8 (11)
Skin Infection (Infections and infestations) | 1 (1)
Eye Infection (Infections and infestations) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary- Other (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Elevated Alkaline phosphatase (Metabolism and nutrition disorders) | 15 (15)
Elevated ALT (Metabolism and nutrition disorders) | 7 (9)
Elevated AST (Metabolism and nutrition disorders) | 7 (10)
Elevated serum bilirubin (Metabolism and nutrition disorders) | 2 (2)
Elevated creatinine (Metabolism and nutrition disorders) | 11 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Low serum bicarbonate (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (10)
Elevated lipase (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (8)
Confusion (Psychiatric disorders) | 4 (4)
Somnolence (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Involuntary movement (Nervous system disorders) | 3 (3)
Sensory neuropathy (Nervous system disorders) | 8 (8)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 8 (10)
Agitation (Psychiatric disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 7 (8)
Flushing (Vascular disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Flu-like syndrome (General disorders) | 3 (3)
Phlebitis (Vascular disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
GI Pain (Gastrointestinal disorders) | 15 (22)
Lung Pain (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 67 (100)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Pelvis pain (Reproductive system and breast disorders) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 2 (2)
Skin pain (Skin and subcutaneous tissue disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Dermatology- Other (Skin and subcutaneous tissue disorders) | 8 (9)
Vascular- Other (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No